CLINICAL TRIAL: NCT06631638
Title: Planned vs. Actual Acetabular Cup Position in Total Hip Arthroplasty With Non-Invasive Navigation
Brief Title: EMPHASYS Cup Positioning in THA With Non-Invasive Navigation (Velys Hip Navigation (VHN))
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSJ202006; DSJ202006 (Other: DePuy Orthopaedics)
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis; Traumatic Arthritis; Rheumatoid Arthritis; Congential Hip Dysplasia; Avascular Necrosis of the Femoral Head; Certain Cases of Ankylosis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Femur Head Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EMPHASYS Cup with VHN (Other): EMPHASYS Cup with Non-Invasive Navigation
  Interventions: Device: EMPHASYS Cup with VHN

INTERVENTIONS:
Device: EMPHASYS Cup with VHN — Total Hip Replacement with EMPHASYS Acetabular shell and Non-Invasive Navigation

SUMMARY:
The purpose of this research is to gather clinical and radiographic (X-ray) information about EMPHASYS™ acetabular shell (also called a hip 'cup') placement in total hip replacement surgery using a non-invasive surgical navigation system called VELYS™ hip navigation system with CUPTIMIZE™ Advanced Hip-Spine Analysis software.

Data collected in this study will be compared with data collected from implantations using different cup positioning instrumentation and techniques to assess performance.

ELIGIBILITY:
Inclusion Criteria:

1. All hip replacement component devices are to be used according to the approved indications.
2. The subject is undergoing a standard of care primary uncemented hip replacement with the EMPHASYS cup and a CORAIL, EMPHASYS or ACTIS stem via the posterolateral, anterolateral, or direct lateral approach with the subject in the lateral decubitus position.
3. The subject is a candidate for implantation utilizing the VELYS Hip Navigation system with CUPTIMIZE advanced
4. Individuals who are able to speak, read, and comprehend the Informed Participant Consent Document and willing and able to provide consent for participation in the study and have authorized the transfer of his/her information to DePuy Synthes.
5. Individuals who are willing and able to complete follow-up as specified by the study protocol.
6. Individuals who are willing and able to complete the Subject Hip Outcomes questionnaires (i.e., FJS-12, EQ-5D-5L and Hip Evaluation) as specified by the study protocol.
7. Individuals who are not bedridden per the discretion of the investigator.
8. Individuals who are a minimum age of 21 years at the time of consent

Exclusion Criteria:

1. Active local or systemic infection.
2. Loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
3. Poor bone quality, such as osteoporosis, where, in the surgeon's opinion, there could be considerable migration of the prosthesis or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the implant(s).
4. Charcot's or Paget's disease.
5. The Subject is a woman who is pregnant or lactating.
6. Subject had a contralateral amputation.
7. Previous partial hip replacement in affected hip.
8. Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three months.
9. Contralateral hip was replaced less than 6 months prior to surgery date.
10. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
11. Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
12. Subject has a medical condition with less than 2 years of life expectancy.
13. Subject, in the opinion of the Investigator, is a drug or alcohol abuser or has a psychological disorder that could affect their ability to complete subject reported questionnaires or be compliant with follow-up requirements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint: Acetabular Cup Position Success at 6 Weeks | 6 Weeks
  For an individual cup position to be considered successful, the cup's placement must satisfy all of the following criteria at 6 weeks: Inclination Success: within 10 degrees of the planned inclination via the surgeon-defined preoperative plan and version Success: within 10 degrees of the planned version via the surgeon-defined preoperative plan.

SECONDARY OUTCOMES:
Inclination Success | 6 weeks
  Inclination Success: within 10 degrees of the planned inclination via the surgeon-defined preoperative plan.
Version Success | 6 weeks
  Version Success: within 10 degrees of the planned version via the surgeon-defined preoperative plan.
Final Intraoperative Inclination | 12 weeks
  Number of participants with final intraoperative inclination will be reported.
Final Intraoperative Version | 12 weeks
  Number of participants with final intraoperative version will be reported.
Harris Hip Score | 12 weeks
  Functional and health status as measured with the Harris Hip Score. This is a validated scoring system of the hip that has a result range of 0-100; the higher the score, the better the patient outcome.
Radiographic Outcomes | 12 weeks
  High quality antero-posterior and lateral radiographs of the operative hip will be obtained during the same intervals as for the clinical evaluations. Views include the Standing AP Hip, Standing AP Pelvis, and Lateral (Modified Lauenstein) Hip. Preoperatively an additional three views will be taken including Lateral flex-seated, Lateral Standing and Standing AP Pelvis.
EQ-5D-5L | 12 weeks
  EuroQol 5D 3L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Forgotten Joint Score | 6 weeks
  Functional and health status as measured with the Forgotten Joint Score (FJS-12). This is a validated score that assesses patient outcomes. The result range is 0-100 where a higher score mean a more favorable result.
Operating Room Times | Immediately after the Surgical Procedure
  Evaluate various operating room times such as anesthesia, fluoroscopy and surgical times.
Leg Length Discrepancy | Immediately after the Surgical Procedure
  Leg Length discrepancy compared to surgeon target based on pre-operative planning
Complication Rates | 30 days
  30-day Complication Rate
Complication Rates | 90 days
  90-day Complication Rate

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UC Davis Health System, Sacramento, California
  - Florida Orthopaedic Institute, Gainesville, Florida
  - Northwell Health, Lake Success, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Orthopaedic and Sports Medicine Center, Gastonia, North Carolina